CLINICAL TRIAL: NCT04319588
Title: Parasternal Block for Postoperative Analgesia in Cardiac Surgery: a Pilot Controlled Trial
Brief Title: Parasternal Block for Cardiac Surgery
Acronym: Parasternal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Giulia Nonnis, Principal Investigator, Campus Bio-Medico University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20/20 PAR ComEt CBM
Record Dates: First submitted 2020-03-09; First posted 2020-03-24 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Cardiac Disease; Analgesia; Acute Pain; Postoperative Pain
MeSH Terms: conditions — Heart Diseases; Agnosia; Acute Pain; Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parasternal Group (Experimental): The "parasternal group" of patients will receive the pre-operative parasternal block (20 ml of 0.5% Ropivacaine per side) in association with infiltration with local anesthetic of access to thoracic drainage (drainage infiltration with 20 ml of 0.25% Ropivacaine) at the end of the intervention combined to General Anesthesia.
  Interventions: Procedure: Parasternal Block+ Infiltration with local anesthetic of access to thoracic drainage
- Case control group (Active Comparator): The "case control group" will only receive drainage infiltration with local anesthetic and standard intraoperative management with opioids.
  Interventions: Procedure: Infiltration with local anesthetic of access to thoracic drainage

INTERVENTIONS:
Procedure: Parasternal Block+ Infiltration with local anesthetic of access to thoracic drainage — After induction of general anesthesia we will perform an ultrasound-guided Parasternal Block in association with infiltration with local anesthetic of access to thoracic drainage at the end of the intervention.
  Arms: Parasternal Group
Procedure: Infiltration with local anesthetic of access to thoracic drainage — Infiltration with local anesthetic of access to thoracic drainage at the end of the intervention.
  Arms: Case control group

SUMMARY:
This study examine the effect of Parasternal Intercostal Nerve Blocks with local anesthetic on pain control in patients undergoing non-emergent cardiac surgery in a prospective controlled trial. Half of participants will receive General Anesthesia combined to parasternal block while the other half receive only General Anesthesia.

DETAILED DESCRIPTION:
60 patients undergoing elective cardiac surgery will be enrolled and divided into two groups:

1. Interventional (parasternal group)
2. Case control group The "parasternal group" of patients will receive the pre-operative parasternal block (20 ml of 0.5% Ropivacaine per side) in association with infiltration with local anesthetic of access to thoracic drainage (drainage infiltration with 20 ml of 0.25% Ropivacaine) at the end of the intervention combined to General Anesthesia.

The "case control group" will only receive drainage infiltration with local anesthetic and standard intraoperative management with opioids.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective cardiac surgery
* Age over 18 years
* ASA I-IV
* Approval by the patient of informed consent

Exclusion Criteria:

* Allergy to local anesthetics
* Puncture site infection
* Lack of signing of informed consent
* Weight <30 Kg
* Age <18 years
* Emergency interventions
* ASA > IV
* Sternal dehiscences
* Dementia (for difficulties in managing weaning from mechanical ventilation and pain)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2020-05-09 (Actual); Study Completion 2020-05-19 (Actual)

PRIMARY OUTCOMES:
Maximum Pain Score | 24 hours
  Postoperative pain assessment using the NRS scale (score from 0 to 10)

SECONDARY OUTCOMES:
Respiratory performance at the TRI-FLOW | 24 hours
  Respiratory performance is assessed by the number of balls raised during inspiration with the TRI-FLOW
Intraoperative opioid administration | 4 hours
  Quantitative evaluation of opioids needed in the intraoperative period
Total opioids consumption | 24 hours
  Number of opioid deliveries (bolus morphine) in the postoperative period
Time to first opioid | 48 hours
  The time in minutes between awakening and the first opioid administration

CONTACTS AND LOCATIONS:
Locations (1):
- Campus Biomedico University, Rome, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chou R, Gordon DB, de Leon-Casasola OA, Rosenberg JM, Bickler S, Brennan T, Carter T, Cassidy CL, Chittenden EH, Degenhardt E, Griffith S, Manworren R, McCarberg B, Montgomery R, Murphy J, Perkal MF, Suresh S, Sluka K, Strassels S, Thirlby R, Viscusi E, Walco GA, Warner L, Weisman SJ, Wu CL. Management of Postoperative Pain: A Clinical Practice Guideline From the American Pain Society, the American Society of Regional Anesthesia and Pain Medicine, and the American Society of Anesthesiologists' Committee on Regional Anesthesia, Executive Committee, and Administrative Council. J Pain. 2016 Feb;17(2):131-57. doi: 10.1016/j.jpain.2015.12.008. PMID 26827847